CLINICAL TRIAL: NCT01926197
Title: A Randomized Phase III Study Evaluating Modified FOLFIRINOX (mFFX) With or Without Stereotactic Body Radiotherapy (SBRT) in the Treatment of Locally Advanced Pancreatic Cancer: A Pancreatic Cancer Radiotherapy Study Group (PanCRS) Trial
Brief Title: Phase 3 Study of FOLFIRINOX (mFFX) +/- SBRT in Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Lucas Kas Vitzthum, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-27492; PANC0015 (Other: OnCore); NCI-2013-01658 (Other: NCI)
Record Dates: First submitted 2013-08-15; First posted 2013-08-20 (Estimated); Results first posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; irinotecan sucrosofate; Leucovorin; Fluorouracil; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified FOLFIRINOX (Active Comparator): Modified FOLFIRINOX (mFFX), a chemotherapeutic treatment regimen of 5FU, leucovorin, irinotecan, and oxaliplatin.
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin; Drug: 5FU
- Modified FOLFIRINOX plus Stereotactic Body Radiotherapy (Experimental): Modified FOLFIRINOX (mFFX), a chemotherapeutic treatment regimen of 5FU, leucovorin, irinotecan, and oxaliplatin, in combination with stereotactic body radiotherapy (SBRT)
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin; Drug: 5FU; Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 85 mg/m² IV over 2 hours on Day 1 of a 14-day cycle.
  Other Names: Eloxatin
Drug: Irinotecan — Irinotecan 180 mg/m² IV over 90 minutes on Day 1 of a 14-day cycle.
  Other Names: Camptosar; Camptothecin-11 (CPT-11); Campto; Onivyde
Drug: Leucovorin — Leucovorin 400 mg/m² IV over 2 hours on Day 1 of a 14-day cycle.
  Other Names: Folinic acid; Wellcovorin; Citrovorum Factor
Drug: 5FU — 5FU 2,400 mg/m² IV over 46 to 48 hours starting on Day 1 of a 14-day cycle.
  Other Names: 5-fluorouracil; Tolak; Fluoroplex; Efudex; Carac; Adrucil
Radiation: Stereotactic Body Radiotherapy (SBRT) — Radiotherapy treatment starting about 8 weeks after modified FOLFIRINOX induction chemotherapy, administered as 5 fractions of 8 Grey (Gy) each, on 5 separate days.
  Arms: Modified FOLFIRINOX plus Stereotactic Body Radiotherapy

SUMMARY:
The goal of this study is to determine the safety and efficacy of a chemotherapy regimen known as Modified FOLFIRINOX (mFFX) alone or with the addition of Stereotactic Body Radiotherapy (SBRT). We hope to learn if this new treatment combination helps to control the disease and improve survival for patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
Primary Objective:

To determine progression free survival for mFFX +/- SBRT.

Secondary Objectives:

* To determine metastasis free survival following mFFX chemotherapy alone or with SBRT.
* To determine the overall survival in pancreatic cancer patients treated with chemotherapy +/- SBRT.
* To determine local progression-free survival in pancreatic cancer patients after chemotherapy +/- SBRT.
* To evaluate acute (within 3 months of treatment) grade 2 or greater gastritis, fistula, enteritis, or ulcer and any other grade 3-4 gastrointestinal toxicity within 3 months of treatment.
* To evaluate the utility of FDG-PET for treatment planning and estimation of progression free survival.
* To identify new biomarkers in pancreatic cancer.
* To evaluate the quality of life of patients before and after either chemotherapy or chemotherapy and SBRT.

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically-confirmed adenocarcinoma of the pancreas
* Determined unresectable by a pancreatic cancer surgeon or a multi-disciplinary or gastrointestinal oncology Tumor Board.
* Stable or better disease on re-staging scans
* Typically, tumors < 8.0 cm in greatest axial dimension but final determination of eligibility based upon radiation normal tissue constraints
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1, or 2
* Leukocytes (white blood cells, WBC) ≥ 3,000/mL
* Absolute neutrophil count (ANC) ≥ 1,500/mL
* Platelets ≥ 50,000/mL
* Total bilirubin ≤ 1.5 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤ 2.5 X institutional ULN
* Creatinine within normal institutional limits
* Ability to understand and the willingness to sign an informed consent form
* Life expectancy > 6 months

EXCLUSION CRITERIA

* Metastatic disease
* Prior radiotherapy to the upper abdomen/liver.
* Prior chemotherapy for pancreatic cancer, other than up to 4 cycles of modified FOLFIRINOX.
* Age < 18 years
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection (or infections requiring systemic antibiotic treatment)
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements.
* Any concurrent malignancy other than non-melanoma skin cancer, non-invasive bladder cancer, or carcinoma in situ of the cervix. Patients with a previous malignancy without evidence of disease for > 5 years will be allowed to enter the trial.
* Pregnant or lactating
* Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control (hormonal or barrier method of birth control; abstinence) for duration of the study
* Women who are not post-menopausal (as defined in Appendix III) and have a positive urine or serum pregnancy test or refuse to take a pregnancy test
* Male subjects who are unwilling or unable to use effective contraception for duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-08-14 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T Chang, Principal Investigator — Stanford University
Locations (9):
- United States (7):
  - UCLA, Los Angeles, California
  - UCSF, San Francisco, California
  - Stanford University, School of Medicine, Stanford, California
  - Loyola University, Maywood, Illinois
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Canada (2):
  - BC Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Modified FOLFIRINOX: Modified FOLFIRINOX (mFFX), a chemotherapeutic treatment regimen of 5FU, leucovorin, irinotecan, and oxaliplatin.
  * Oxaliplatin 85 mg/m² IV over 2 hours on Day 1 of a 14-day cycle.
  * Irinotecan 180 mg/m² IV over 90 minutes on Day 1 of a 14-day cycle.
  * Leucovorin 400 mg/m² IV over 2 hours on Day 1 of a 14-day cycle.
  * 5FU: 5FU 2,400 mg/m² IV over 46 to 48 hours starting on Day 1 of a 14-day cycle.
- Modified FOLFIRINOX Plus Stereotactic Body Radiotherapy: Modified FOLFIRINOX (mFFX), a chemotherapeutic treatment regimen of 5FU, leucovorin, irinotecan, and oxaliplatin, in combination with stereotactic body radiotherapy (SBRT)
  * Oxaliplatin 85 mg/m² IV over 2 hours on Day 1 of a 14-day cycle.
  * Irinotecan 180 mg/m² IV over 90 minutes on Day 1 of a 14-day cycle.
  * Leucovorin 400 mg/m² IV over 2 hours on Day 1 of a 14-day cycle.
  * 5FU: 5FU 2,400 mg/m² IV over 46 to 48 hours starting on Day 1 of a 14-day cycle.
  * Stereotactic Body Radiotherapy (SBRT): Radiotherapy treatment starting about 8 weeks after modified FOLFIRINOX induction chemotherapy, administered as 5 fractions of 8 Grey (Gy) each, on 5 separate days.
Period: Overall Study
Arm/Group | Modified FOLFIRINOX | Modified FOLFIRINOX Plus Stereotactic Body Radiotherapy
Started | 13 | 14
Completed | 12 | 13
Not Completed | 1 | 1
Not completed — Withdrawn to receive chemotherapy | 1 | 0
Not completed — Withdrawn due to non-coverage by insurance | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only participants that received study treatment are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified FOLFIRINOX | Modified FOLFIRINOX Plus Stereotactic Body Radiotherapy | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 6 | 5 | 11
Age, Continuous [Median (Standard Deviation); unit: years] | 64.1 (8.0) | 62.0 (7.3) | 63 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 3 | 9 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 10 | 12 | 22
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) means the period of time that a participant remains alive without tumor progression either locally or at a distant site in the body (metastasis). The effect of the study treatments was assessed as the median PFS of participants in the treatment groups. The outcome is reported as the median PFS with standard deviation.
Time Frame: 38 months
Measure: Median (Standard Deviation); unit: months
Arm/Group | Modified FOLFIRINOX | Modified FOLFIRINOX Plus Stereotactic Body Radiotherapy
Number analyzed (Participants) | 13 | 12
months | 6.5 (6.6) | 8.4 (9.5)

2. Secondary Outcome: Local Progression-free Survival (Local PFS)
Description: Local progression-free survival (PFS) means the period of time that a participant remains alive without recurrence or advancement of the disease at the baseline sites of the tumor (local progression). The effect of the study treatments was assessed as the median local PFS of participants in the treatment groups. The outcome is reported as the median local PFS with standard deviation.
Time Frame: 38 months
Measure: Median (Standard Deviation); unit: months
Arm/Group | Modified FOLFIRINOX | Modified FOLFIRINOX Plus Stereotactic Body Radiotherapy
Number analyzed (Participants) | 13 | 12
months | 6.5 (6.6) | 8.4 (10.5)

3. Secondary Outcome: Progression-free Survival (PFS) at 1 Year
Description: Progression-free survival (PFS) means the period of time that a participant remains alive without tumor progression either locally or at a distant site in the body (metastasis). The effect of the study treatments was assessed as the number of participants in each treatment group that remained alive without tumor progression, at 1 year after treatment.
  The outcome is reported as a number without dispersion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Modified FOLFIRINOX | Modified FOLFIRINOX Plus Stereotactic Body Radiotherapy
Number analyzed (Participants) | 13 | 12
Participants | 5 | 2

4. Secondary Outcome: Metastasis-free Survival (MFS)
Description: Metastasis-free survival (MFS) means the period of time that a participant remains alive without the appearance of new tumor lesions a distant site in the body (metastasis). The effect of the study treatments was assessed as the median MFS of participants in the treatment groups. The outcome is reported as the median PFS with standard deviation.
Time Frame: 62 months
Measure: Median (Standard Deviation); unit: months
Arm/Group | Modified FOLFIRINOX | Modified FOLFIRINOX Plus Stereotactic Body Radiotherapy
Number analyzed (Participants) | 13 | 12
months | 12.9 (6.4) | 10.8 (16.9)

5. Secondary Outcome: Overall Survival (OS)
Description: The effect of the study treatments was assessed as the length of time participants in each treatment group that remained alive. The outcome is reported as the median OS with standard deviation.
Time Frame: 62 months
Measure: Median (Standard Deviation); unit: months
Arm/Group | Modified FOLFIRINOX | Modified FOLFIRINOX Plus Stereotactic Body Radiotherapy
Number analyzed (Participants) | 13 | 12
months | 12.9 (6.4) | 13.4 (16.6)

6. Secondary Outcome: Grade 2 or Greater Gastrointestinal (GI) Toxicity
Description: Toxicity means an adverse event related to the study treatment. Toxicity was assessed between treatment groups as the number of treatment-related , ≥ grade 2 events of gastritis, fistula, enteritis, or ulcer; plus any other Grade 3 to 5 gastrointestinal (GI) toxicity. The outcome is reported as the number of defined adverse events by preferred term for each treatment group, occurring within 3 months of the start of treatment. These adverse events by definition are all within the Common Terminology Criteria for Adverse Events (CTCAE) version 4.01 Gastrointestinal Body System. The outcome is reported as numbers without dispersion.
  All-cause Mortality mFFX 7 SBRT 8
Time Frame: 3 months
Population: Analysis group is those participants that received at least one dose of the Modified FOLFIRINOX (mFFX) chemotherapy regimen.
Measure: Number; unit: Related adverse events
Arm/Group | Modified FOLFIRINOX | Modified FOLFIRINOX Plus Stereotactic Body Radiotherapy
Number analyzed (Participants) | 13 | 12
Related adverse events
  Blood in stool (melena) | 1 | 0
  Colitis | 1 | 0
  Colonic obstruction | 1 | 0
  Diarrhea | 3 | 0
  Duodenal perforation | 0 | 1
  Fistula, anal | 0 | 3
  Fluid in abdomen (ascites) | 0 | 2
  Gastrointestinal bleed (hemorrhage) | 1 | 1
  Gastrointestinal bleed (hemorrhage), upper | 0 | 3
  Gastrointestinal inflammation (enterocolitis) | 1 | 0
  Nausea | 3 | 1
  Pain, abdominal | 3 | 4
  Pain, intractable (due to disease progression) | 0 | 1
  Stool discolored, clay color | 1 | 0
  Vomited blood (hematemesis) | 0 | 4

ADVERSE EVENTS:
Time Frame: up to 62 months
Arm/Group | Modified FOLFIRINOX | Modified FOLFIRINOX Plus Stereotactic Body Radiotherapy
All-Cause Mortality (participants affected / at risk) | 7/12 | 8/13
Serious Adverse Events (participants affected / at risk) | 5/12 | 7/13
Other Adverse Events (participants affected / at risk) | 12/12 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified FOLFIRINOX (N=12) | Modified FOLFIRINOX Plus Stereotactic Body Radiotherapy (N=13)
Other, hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bleed (hemorrhage), gastrointestinal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bleed (hemorrhage), gastrointestinal upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pain, intractable (due to disease progression) (General disorders) | 0 (0) | 1 (1)
Lung infection - Klebsiella pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Other, renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified FOLFIRINOX (N=12) | Modified FOLFIRINOX Plus Stereotactic Body Radiotherapy (N=13)
Anemia (Blood and lymphatic system disorders) | 10 (88) | 11 (100)
White blood cell (WBC) count elevated (leukocytosis) (Blood and lymphatic system disorders) | 5 (20) | 7 (15)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ringing in the ears (tinnitus) (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Eye inflammation (scleral disorder) (Eye disorders) | 0 (0) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abnormal sensation in the mouth (oral dysesthesia) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 2 (5)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (4)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Anemia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Bleed (hemorrhage), gastrointestinal upper (Gastrointestinal disorders) | 0 (0) | 1 (3)
Bloating (Gastrointestinal disorders) | 4 (7) | 4 (11)
Constipation (Gastrointestinal disorders) | 3 (19) | 7 (23)
Diarrhea (Gastrointestinal disorders) | 11 (36) | 6 (36)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (3) | 2 (5)
Fluid in abdomen (ascites) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, anal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, hemorrhoidal (Gastrointestinal disorders) | 0 (0) | 1 (8)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (5)
Indigestion (dyspepsia) (Gastrointestinal disorders) | 2 (5) | 3 (4)
Inflammation of the lining of the stomach (gastritis) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (38) | 9 (57)
Oral inflammation (mucositis) (Gastrointestinal disorders) | 2 (4) | 3 (5)
Other, excess in the stool (steatorrhea) (Gastrointestinal disorders) | 1 (3) | 0 (0)
Other, stool discolored, clay color (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain, abdominal (Gastrointestinal disorders) | 9 (22) | 10 (37)
Pain, rectal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain, stomach (Gastrointestinal disorders) | 1 (2) | 0 (0)
Swallowing difficulty (dysphagia) (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (6) | 4 (19)
Chills (General disorders) | 1 (1) | 3 (5)
Edema, localized (General disorders) | 1 (2) | 0 (0)
Edema, peripheral (General disorders) | 4 (8) | 1 (1)
Fatigue (General disorders) | 12 (63) | 10 (55)
Fever (General disorders) | 1 (1) | 2 (2)
Flu-like symptoms (General disorders) | 1 (1) | 2 (6)
General feeling of discomfort (malaise) (General disorders) | 2 (2) | 2 (2)
Infusion-related reaction (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 3 (15) | 5 (9)
Pain, abdominal (General disorders) | 1 (1) | 1 (1)
Pain, chest, non-cardiac (General disorders) | 1 (2) | 1 (1)
Clot in portal vein (thrombosis) (Hepatobiliary disorders) | 0 (0) | 1 (5)
Platelet count decreased (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (2) | 2 (2)
Rash, papulopustular (Infections and infestations) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (3)
Alanine aminotransferase increased (Investigations) | 6 (22) | 5 (9)
Alkaline phosphatase decreased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 10 (43) | 9 (44)
Aspartate aminotransferase increased (Investigations) | 12 (20) | 2 (4)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0)
Cardiac troponin increased (Investigations) | 0 (0) | 1 (2)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyl transferase (GGT) increased (Investigations) | 1 (2) | 0 (0)
International normalized ratio (INR) increased (Investigations) | 0 (0) | 1 (4)
Leukocytosis (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (13) | 8 (38)
Lymphocyte count increased (Investigations) | 1 (2) | 3 (4)
Neutrophil count decreased (Investigations) | 2 (5) | 3 (8)
Other, Creatinine decreased (Investigations) | 1 (1) | 0 (0)
Other, Neutrophil count increase (Investigations) | 1 (1) | 0 (0)
Other, Protein total decrease (Investigations) | 1 (1) | 0 (0)
Other, WBC morphology (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 11 (61) | 9 (55)
Protein total decreased (Investigations) | 0 (0) | 1 (1)
Reduced red blood cells or hemoglobin (anemia) (Investigations) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 1 (2) | 1 (1)
Weight loss (Investigations) | 10 (39) | 4 (42)
White blood cell decreased (Investigations) | 6 (13) | 5 (15)
Decreased appetite (anorexia) (Metabolism and nutrition disorders) | 8 (29) | 4 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (27) | 10 (74)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (24) | 9 (64)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (13) | 6 (29)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 7 (15) | 5 (17)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5) | 6 (14)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Other, Phosphate increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (5) | 2 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3)
Muscle pain (myalgia) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain, back (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (17)
Pain, flank (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Anxiety (Nervous system disorders) | 1 (2) | 0 (0)
Bad taste in mouth (dysgeusia) (Nervous system disorders) | 3 (8) | 1 (2)
Depression (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Drowsiness, unusual (somnolence) (Nervous system disorders) | 1 (11) | 1 (1)
Excessive sleep (hypersomnia) (Nervous system disorders) | 0 (0) | 1 (1)
Feeling faint (presyncope) (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Movements involuntary (Nervous system disorders) | 1 (2) | 0 (0)
Nerve damage or injury (neuropathy) (Nervous system disorders) | 7 (40) | 8 (29)
Nerve damage or injury (neuropathy), peripheral (Nervous system disorders) | 0 (0) | 3 (6)
Nerve damage or injury (neuropathy), peripheral sensory (Nervous system disorders) | 1 (1) | 0 (0)
Nerve tingling (paresthesia) (Nervous system disorders) | 1 (2) | 2 (3)
Nosebleed (epistaxis) (Nervous system disorders) | 0 (0) | 1 (1)
Other, muscle weakness (Nervous system disorders) | 0 (0) | 1 (1)
Other, tremor (Nervous system disorders) | 0 (0) | 1 (1)
Reduced albumin in the blood (hypoalbuminemia) (Nervous system disorders) | 0 (0) | 1 (1)
Slow or slurred speech (dysarthria) (Nervous system disorders) | 1 (1) | 0 (0)
Tiredness (fatigue) (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Amnesia (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (5) | 3 (15)
Confusion (Psychiatric disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (5) | 3 (4)
Difficulty sleeping (insomnia) (Psychiatric disorders) | 2 (2) | 2 (13)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (3)
Excess protein in urine (proteinuria) (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (7)
Urinary urgency (Renal and urinary disorders) | 1 (2) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 1 (1)
Edema, pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Labored breathing (dyspnea) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Lung collaspe (atelectasis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (7)
Excessive sweating (hyperhidrosis) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hair loss, immune-realted (alopecia) (Skin and subcutaneous tissue disorders) | 2 (10) | 0 (0)
Itch (pruritus) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Other, atypical junctional nevus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other, axilla boil (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Other, aypical melanocytic proliferation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other, bump on right upper extremity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other, deep mobile mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other, medial right nodule on right upper extremity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other, melanoma in-situ (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other, small nodule on right upper extremity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (6) | 0 (0)
Rash, maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Edema (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 8 (32) | 8 (27)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT01926197/Prot_SAP_001.pdf
  • Informed Consent Form (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT01926197/ICF_000.pdf